CLINICAL TRIAL: NCT02985437
Title: Safety and Tolerability of Topically Applied Bovine Lung Surfactant on Intact Skin and Superficial Subepidermal Lesions in Healthy Volunteers
Brief Title: Safety and Tolerability of Topically Applied Bovine Lung Surfactant on Intact Skin
Acronym: SATOSU
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Prof. Dr. Dr. Ursula Mirastschijski (Other)
Collaborators: European Research Council (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Dr. Ursula Mirastschijski, Principal Investigator, University of Bremen
Organization: University of Bremen (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMWH01; 2015-000890-11 (EudraCT Number); DRKS00011353 (Other: German Clinical Trials Register (DRKS))
Record Dates: First submitted 2016-11-28; First posted 2016-12-07 (Estimated); Last update posted 2017-09-07 (Actual); Status verified 2017-09

CONDITIONS: Skin and Connective Tissue Diseases
Keywords: wound healing; Bovine Lung Surfactant; SATOSU
MeSH Terms: conditions — Skin and Connective Tissue Diseases | interventions — Surface-Active Agents; Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Surfactant (Experimental): Alveofact® (Bovine Lung Surfactant), 0.5 mg/ml per day (solution) all two days maximal eight times
  Interventions: Drug: Surfactants
- Saline (Active Comparator): 0.9% Sodium chloride solution (NaCl solution), 2 ml per day (solution) all two days maximal eight times
  Interventions: Drug: Saline Solution

INTERVENTIONS:
Drug: Surfactants
  Arms: Surfactant
Drug: Saline Solution
  Arms: Saline

SUMMARY:
Bovine Lung Surfactant is used as standard therapy for reducing alveolar surface tension in preterm infants. Here the drug is administered via airways.

The use on skin to stimulate the wound healing has not yet been tested in humans, i.e. it is not yet approved for the treatment of wound healing disorders. In the planned clinical trial Lung Surfactant is used the first time for the local treatment of skin lesions in humans. No substance related side effects were observed during the application via airways in neonates.

The innovative idea to use lung surfactant for skin wound healing derived from two observations. First, when the skin is injured, the barrier protecting the moist body surface from the dry environment is discontinued and in part lost.

Lung surfactant has several characteristics that might be beneficial for treatment of chronic cutaneous wounds.

ELIGIBILITY:
Inclusion Criteria:

* Two healthy forearms,
* No known chronical skin diseases,
* Dermatoses or allergies,
* Signed form of consent,
* Caucasian

Exclusion Criteria:

* Pregnancy or nursing period,
* Diabetes (Type I or II),
* Systemic or infectious diseases,
* Skin disease,
* Known allergies against bovine products or wound dressings,
* Mental diseases, missing ability to consent,
* Addictive disorders (e.g. alcohol, drugs),
* Peripheral circulatory disorder, Morbus Raynaud,
* Current (or < 4 weeks ago) participation in clinical trials

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-12-08 (Actual); Primary Completion 2017-08-30 (Actual); Study Completion 2017-08-30 (Actual)

PRIMARY OUTCOMES:
Tolerability of Lung Surfactant in cutaneous application measured by mean Clinical Scoring Scale for dermatitis (CSS) computed over all visits | days 2,4,6,8,10,12,14 post baseline

SECONDARY OUTCOMES:
Time to wound conclusion of wound healing and reepithelialisation: measurement of wound surface | up to 14 days and one time follow up after 30 days
Pain measured by mean Visual Analogue Scale over all visits | days 2,4,6,8,10,12,14 post baseline
TransEpidermal Water Loss = indirect measurement of reepithelialisation and of wound closure | day 2
TransEpidermal Water Loss = indirect measurement of reepithelialisation and of wound closure | day 4
TransEpidermal Water Loss = indirect measurement of reepithelialisation and of wound closure | day 6
TransEpidermal Water Loss = indirect measurement of reepithelialisation and of wound closure | day 8
TransEpidermal Water Loss = indirect measurement of reepithelialisation and of wound closure | day 10
TransEpidermal Water Loss = indirect measurement of reepithelialisation and of wound closure | day 12
TransEpidermal Water Loss = indirect measurement of reepithelialisation and of wound closure | day 14

OTHER OUTCOMES:
Adverse Events | up to 14 days and one time follow up after 30 days
Number of Participants With Abnormal Laboratory Values | Baseline and day 14

CONTACTS AND LOCATIONS:
Overall Officials: Ursula Mirastschijski, Prof. Dr., Principal Investigator — University of Bremen
Locations (1):
- University of Bremen, Bremen, Germany

IPD SHARING:
Plan to Share IPD: No